CLINICAL TRIAL: NCT02856464
Title: A Phase II Prospective Trial of Prophylactic Donor Lymphocyte Infusions for the Prevention of Relapse Post HSCT in Patients With High Risk Myeloid Malignancy
Brief Title: Prophylactic DLI for the Prevention of Relapse Post HSCT in Patients With High Risk Myeloid Malignancy
Acronym: PRO-DLI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-DLI
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: DLI will be administered to all patients at Month 4 (+/- 20 days) after stem cell transplant regardless of peripheral blood CD3 chimerism (including if they have full donor chimerism)
- Control (Other)
  Interventions: Other: DLI will be administered from Month 6 (+/- 20 days) after stem cell transplant according to institutional practice

INTERVENTIONS:
Other: DLI will be administered to all patients at Month 4 (+/- 20 days) after stem cell transplant regardless of peripheral blood CD3 chimerism (including if they have full donor chimerism)
  Arms: Experimental
Other: DLI will be administered from Month 6 (+/- 20 days) after stem cell transplant according to institutional practice
  Arms: Control

SUMMARY:
The trial will be conducted as a multicentre open label, randomised prospective phase II clinical trial in patients with high risk myeloid malignancies.

The primary objective is to evaluate whether prophylactic donor lymphocyte infusions (DLI) delivered as part of a planned schedule improves the disease free survival of patients with myeloid malignancies.

ELIGIBILITY:
Patient Inclusion Criteria

1. Haematological cancer which can be one of the following

   1. Acute Myeloid Leukaemia (AML) if Intermediate or High risk in CR1
   2. AML if favourable risk in CR2
   3. Patients with AML or MDS with residual cytogenetic or molecular disease pre-HSCT
   4. CMML
   5. Myelodysplastic Syndrome (MDS) defined by an IPSS category int-1 or higher with <5% blasts at the time of randomisation following cyto-reduction if necessary
   6. Secondary MDS or AML; defined as arising from antecedent haematological disease or secondary to prior chemotherapy.
2. Patients with sibling or 9/10 or 10/10 HLA matched unrelated donor
3. Patients receiving alemtuzumab based reduced intensity conditioned HSCT
4. Age >/=18 years
5. Able to comprehend and give informed consent

Patient Exclusion Criteria

1. Patients with >5% blasts at time of HSCT
2. Patients eligible for myeloablative (Bu/Cy of Cy/TBI) HSCT protocols
3. Patients with myelofibrosis
4. Patients with hypersensitivity to alemtuzumab, melphalan, fludarabine or busulphan
5. ECOG performance status > 2
6. Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | One year

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom